CLINICAL TRIAL: NCT01552551
Title: Assessment and Referral Versus Exercise in Primary Prevention of Falls: PA Healthy Steps Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Steven M. Albert, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: U48DP002657-RCT; U48DP002657 (NIH)
Record Dates: First submitted 2012-03-08; First posted 2012-03-13 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Lower Extremity Weakness Distal; Distorted; Balance
Keywords: Falls; exercise; safety; injury; Older adults
MeSH Terms: conditions — Motor Activity; Wounds and Injuries | interventions — Restraint, Physical; Educational Status; Motion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Healthy Steps (Active Comparator): Healthy Steps program as currently implemented by the PA Department of Aging
  Interventions: Behavioral: Assessment and education
- Healthy Steps with Falls Case Management (Experimental): Healthy Steps program augmented with research interventionist guidance on seeking physician care and home safety assessment
  Interventions: Behavioral: Healthy Steps with Falls Case Management
- Healthy Steps in Motion (Experimental): Healthy Steps program augmented with Healthy Steps in Motion, a 4-week, twice a week program of group exercise.
  Interventions: Behavioral: Healthy Steps in Motion

INTERVENTIONS:
Behavioral: Assessment and education — PA Healthy Steps program
  Arms: Healthy Steps
Behavioral: Healthy Steps with Falls Case Management — Counseling to ensure that participants receive a physician assessment and home safety check
  Arms: Healthy Steps with Falls Case Management
Behavioral: Healthy Steps in Motion — Group exercise program
  Arms: Healthy Steps in Motion

SUMMARY:
Older adults at high risk of falls will complete the PA Healthy Steps program. This program will be implemented by research staff who will follow the training manual and implement the program as it was designed to assess the effectiveness of the program. Participants will then be randomly assigned to three arms: (i) Follow-up only; (ii) Falls case management, in which adherence to physician and home safety assessments will be facilitated; and (iii) Healthy Steps in Motion, a 4-week group exercise program designed to complement Healthy Steps. All participants will be followed monthly for 6 months through personal and automated telephone interview protocols to ascertain falls and injuries.

DETAILED DESCRIPTION:
This falls prevention program is offered in 11 senior housing sites. Trained instructors from the research team provide the Healthy Steps in Motion exercise classes. Participants provide a signed form indicating physician clearance for participation. Falls case management involves monthly calls to speak with participants about home safety checks, perceived risk for falls, and physician contact or other visits to health care professionals to reduce falls risk.

This study is a pilot. The research team is interested in participation and adherence, as well as the primary outcome of falls incidence.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent
2. Willing to be randomized
3. Scoring in the lowest tertile on at least one test in the Healthy Steps lower extremity performance battery
4. Age 50+

Exclusion Criteria:

1. Hospice enrollee or life-threatening illness
2. Active cancer treatment
3. Neurologic disease linked to falls risk, such as Parkinson's
4. Unable to ambulate indoors
5. High likelihood of moving in next 6 months

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2012-05; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Falls | 6 months
  Falls ascertained in automated monthly telephone contact

SECONDARY OUTCOMES:
Fall-related injuries requiring hospitalization/emergency department care | 6 months
  Events ascertained in a monthly automated telephone interview

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Albert, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified research data will be made available to qualified investigators